CLINICAL TRIAL: NCT02111577
Title: A Randomized, Double Blind, Multicenter, Parallel-group, Phase III Study to Evaluate Efficacy and Safety of DCVAC/PCa Versus Placebo in Men With Metastatic Castration Resistant Prostate Cancer Eligible for 1st Line Chemotherapy
Brief Title: Phase III Study of DCVAC/PCa Added to Standard Chemotherapy for Men With Metastatic Castration Resistant Prostate Cancer
Acronym: VIABLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SOTIO a.s. (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP005; 2012-002814-38 (EudraCT Number)
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Immunotherapy; Metastatic; Castration-resistant; Prostate cancer; Biological; Vaccine
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DCVAC/PCa with standard of care chemotherapy (Experimental): Combination therapy with DCVAC/PCa and standard of care chemotherapy (docetaxel and prednisone)
  Interventions: Biological: DCVAC/PCa
- Placebo with standard of care chemotherapy (Placebo Comparator): Combination therapy with placebo and standard of care chemotherapy (docetaxel and prednisone) as comparator
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: DCVAC/PCa — DCVAC/PCa concurrently with docetaxel plus prednisone every 3 weeks (± 7 days). DCVAC/PCa was administered at least 7 days before or and at least 7 days after the nearest chemotherapy (days 8-15 of chemotherapy cycles). After discontinuation of chemotherapy for any reason, each following dose of DCVAC/PCa was given every 4 weeks (-7/+14 days) for up to a total of 15 doses.
  Other Names: Stapuldencel
  Arms: DCVAC/PCa with standard of care chemotherapy
Biological: Placebo — Placebo concurrently with docetaxel plus prednisone every 3 weeks (± 7 days). Placebo was administered at least 7 days before or and at least 7 days after the nearest chemotherapy (days 8-15 of chemotherapy cycles). After discontinuation of chemotherapy for any reason, each following dose of placebo was given every 4 weeks (-7/+14 days) for up to a total of 15 doses.
  Arms: Placebo with standard of care chemotherapy

SUMMARY:
The VIABLE study sought to confirm the hypothesis that the combination of docetaxel with DCVAC/PCa followed by a maintenance therapy with DCVAC/PCa would improve overall survival in patients with metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
This was a randomized, double blind, placebo-controlled, multicenter, international, parallel-group phase III study. Patients with metastatic castration-resistant prostate cancer who were candidates to receive standard of care first-line chemotherapy with docetaxel plus prednisone were randomized 2:1 into one of two arms: an investigational arm (DCVAC/PCa) and a control arm (placebo) in addition to chemotherapy (docetaxel plus prednisone).

ELIGIBILITY:
Inclusion criteria:

* Male 18 years and older.
* Histologically or cytologically confirmed prostate adenocarcinoma.
* Presence of skeletal, or soft-tissue/visceral/nodal metastases according to one of the following criteria:

  * Confirmed pathological fracture related to the disease OR
  * Confirmation of distant bone and/or soft-tissue and/or visceral metastases on CT or MRI scan or bone scintigraphy OR
  * Positive pathology report of metastatic lesion
* Disease progression despite androgen-deprivation therapy (ADT) as indicated by:

  * Prostate-specific antigen (PSA) increase that is ≥ 2 ng/mL and ≥ 25% above the minimum PSA as reached during ADT or above the pre-treatment level, if no response was observed and which is confirmed by a second value 1 or more weeks later OR
  * Progression of measurable lymph nodes (short axis ≥ 15 mm) or visceral lesion measurable per RECIST v1.1 criteria, confirmation by an independent review facility (IRF) required OR
  * Two or more new lesions appearing on bone scan/imaging compared with a previous scan (confirmation by IRF required)
* Maintenance of castrate conditions: patients, who have not had a surgical orchiectomy, must continue with hormone therapy with gonadotropin releasing hormone/ luteinizing hormone-releasing hormone (GnRH/LHRH) agonists or antagonists to reach levels of serum testosterone of ≤ 1.7 nmol/L (50 ng/dL). The duration of the castration period must be at least 4 months before screening as evidenced by combination of clinical/laboratory data (see section 6.8.1).
* Laboratory criteria:

  * White blood cells (WBC) greater than 4,000/mm3 (4.0 x109/L)
  * Neutrophil count greater than 1,500/mm3 (1.5 x109/L).
  * Hemoglobin of at least 10 g/dL (100 g/L).
  * Platelet count of at least 100,000/mm3 (100 x 109/L).
  * Total bilirubin within normal limits (benign hereditary hyperbilirubinemias, e.g. Gilbert's syndrome, are permitted).
  * Serum alanine aminotransferase, aspartate aminotransferase, and creatinine < 1.5x times the upper limit of normal (ULN).
* Life expectancy of at least 6 months based on Investigator's judgment.
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2.
* At least 4 weeks after surgery or radiotherapy before randomization.
* A minimum of 28 days beyond initiation of bisphosphonate or denosumab therapy before randomization.
* Recovery from primary local surgical treatment, radiotherapy or orchiectomy before randomization.
* Signed informed consent including patient's ability to comprehend its contents.

Exclusion criteria:

* Confirmed brain and/or leptomeningeal metastases (other visceral metastases are acceptable).
* Current symptomatic spinal cord compression requiring surgery or radiation therapy.
* Prior chemotherapy for prostate cancer.
* Patient co-morbidities:

  * Subjects who are not indicated for chemotherapy treatment with first line Standard of Care chemotherapy (docetaxel and prednisone).
  * HIV positive, human T-lymphotropic virus positive.
  * Active hepatitis B (active hepatitis B), active hepatitis C (HCV), active syphilis.
  * Evidence of active bacterial, viral or fungal infection requiring systemic treatment.
  * Clinically significant cardiovascular disease including:

    * symptomatic congestive heart failure.
    * unstable angina pectoris.
    * serious cardiac arrhythmia requiring medication.
    * uncontrolled hypertension.
    * myocardial infarction or ventricular arrhythmia or stroke within a 6 months before screening, known left ventricular ejection fraction (LVEF) < 40% or serious cardiac conduction system disorders, if a pacemaker is not present.
  * Pleural and pericardial effusion of any NCI CTCAE grade.
  * Peripheral neuropathy having a NCI CTCAE ≥ grade 2.
  * History of malignant disease (with the exception of non-melanoma skin tumors) in the preceding five years.
  * Active autoimmune disease requiring treatment.
  * History of severe forms of primary immune deficiencies.
  * History of anaphylaxis or other serious reaction following vaccination.
  * Known hypersensitivity to any constituent of the DCVAC/PCa or placebo product.
  * Uncontrolled co-morbidities including, psychiatric or social conditions which, in the Investigator's opinion, would prevent participation in the trial.
* Systemic corticosteroids at doses greater than 40 mg hydrocortisone daily or equivalent for any reason other than treatment of PCa within 6 months before randomization.
* Ongoing systemic immunosuppressive therapy for any reason.
* Treatment with anti-androgens, inhibitors of adrenal-produced androgens or other hormonal tumor-focused treatment performed on the day of randomization (except for GnRH/LHRH agonists or antagonists) to exclude possible anti-androgen withdrawal response. This criterion is not applicable to subjects who have never responded to anti-androgen treatment, as there is no risk of anti-androgen withdrawal response.
* Treatment with immunotherapy against PCa within 6 months before randomization.
* Treatment with radiopharmaceutical within 8 weeks before randomization.
* Participation in a clinical trial using non-immunological experimental therapy within 4 weeks before randomization.
* Participation in a clinical trial using immunological experimental therapy (e.g., monoclonal antibodies, cytokines or active cellular immunotherapies) within 6 months before randomization.
* Refusal to sign the informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1182 (Actual)
Dates: Start 2014-05-26 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J. Vogelzang, Principal Investigator — US Oncology Research/Comprehensive Cancer Centers of Nevada
Locations (177):
- United States (58):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Compassionate Care Research Group, Inc., Corona, California
  - California Cancer Associates for Research and Excellence, Encinitas, California
  - Compassionate Care Research Group, Inc., Fountain Valley, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Hao Wei Zhang, MD, LLC, Los Angeles, California
  - Desert Hematology Oncology Medical Group, Rancho Mirage, California
  - Compassionate Care Research Group, Inc., Riverside, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Oncology Institute of Hope and Innovation, Whittier, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - University of Colorado, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Eastern CT Hematology and Oncololgy Associates, Norwich, Connecticut
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Univ. of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Saint Luke's Cancer Institute, Kansas City, Kansas
  - University of Kansas Cancer Center & Medical Pavilion, Westwood, Kansas
  - Tulane University, New Orleans, Louisiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Associates In Oncology/Hematology,P.C, Rockville, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Umass Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - GU Research Network, Omaha, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Research Centers of Nevada, Henderson, Nevada
  - New Jersey Hematology Oncology Associates, Brick, New Jersey
  - Premier Urology Associates, LLC / AdvanceMed Research, Lawrenceville, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - UC Health University of Cincinnati, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Northwest Cancer Specialists, P.C., Tualatin, Oregon
  - Urologic Consultants of Southeastern Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Cancer Care Associates St. Luke's University and Health Network, Easton, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Associates in Oncology & Hematology, Chattanooga, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - UT Health, Internal Medicine, Division of Oncology, Houston, Texas
  - Texas Health Physicians Group, Plano, Texas
  - Cancer Care Network of South Texas, San Antonio, Texas
  - Tyler Hematology Oncology, Tyler, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - West Virginia University Mary Babb Randolph Cancer Center, Morgantown, West Virginia
- Austria (3):
  - Universitatsklinikum fur Urologie und Andrologie, Salzburg
  - Krankenhaus Barmherzige Brueder, Vienna
  - AKH Universitatskrankenhaus Wien, Vienna
- Belarus (2):
  - N.N. Alexandrov National Research Center, Lesnoy
  - Minsk City Oncological Hospital, Minsk
- Belgium (5):
  - Clinique d'Oncologie Medicale Institut Jules Bordet, Brussels
  - Erasme Hospital- Urologie, Brussels
  - Cliniques Universitaires Saint Luc- Urologie, Brussels
  - Urologie UZ Gent, Ghent
  - Urology Department St. Elizabeth Ziekenhuis, Turnhout
- Bulgaria (5):
  - Specialized Hospital for Active treatment in Oncology, Haskovo
  - Central Oncology Hospital, Plovdiv
  - Complex Oncology Center, Plovdiv
  - Multifunctional Hospital for Active Treatment Serdika, Sofia
  - Specialized Hospital for Active Treatment of Oncology Diseases, Sofia
- Croatia (3):
  - General Hospital Varazdin, Varaždin
  - Clinical Hospital Center Zagreb, Zagreb
  - University Hospital Center Sisters of Charity, Zagreb
- Czechia (11):
  - Onkologicke centrum, Nemocnice Chomutov, Chomutov
  - Klinika onkologie a radioterapie, Fakultni nemocnice, Hradec Králové
  - Nemocnice Jihlava, urologicke oddeleni, Jihlava
  - Urologicke oddeleni, Krajska nemocnice, Liberec
  - Onkologicka klinika, Fakultni nemocnice, Olomouc
  - Klinika onkologicka, Fakultni nemocnice, Ostrava-Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Thomayerova nemocnice, Prague
  - Fakultni nemocnice v Motole, Prague
  - Krajska zdravotni, urologicke oddeleni, Ústí nad Labem
- Rigshospitalet, Copenhagen, Denmark
- France (6):
  - St-Louis IDF Medical Oncology, Paris
  - Hopital St. Joseph, Paris
  - Hospital Cochin, Service de Urologie, Paris
  - HEGP medical oncology, Paris
  - HIA Begin, Saint-Mandé
  - Hospital Civil de Strasbourg, Strasbourg
- Germany (19):
  - Charite Universitatsklinikum Berlin, Berlin
  - Stadtisches Klinikum Braunschweig, Braunschweig
  - Klinik und Poliklinik Urologie, Cologne
  - Universtatsklinikum Carl Gustav Carus, Dresden
  - Waldkrankenhaus St. Marien, Erlangen
  - Krankenhaus Nordwest, Frankfurt
  - Universitatsklinikum Halle (Saale), Halle
  - Asklepios-Klinik Hamburg-Altona, Hamburg
  - Vinzenkrankenhaus Hannover, Hanover
  - Medizinische hochschule Hannover, Hanover
  - Universitatskinikum Jena, Jena
  - Universitatsmedizin Mannheim, Mannheim
  - Universtatsklinikum Munster, Münster
  - Studienpraxis Urologie, Nürtingen
  - Klinikum Oldenburg AOR, Oldenburg
  - Universitastsklinikum Tubingen, Tübingen
  - Universitatsklinikum Ulm, Ulm
  - Ammerland Klinik fur Urologie, Westerstede
  - Praxigemeinschaft fur Onkologie und Urologie, Wilhelmshaven
- Hungary (4):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Egyesitett Szent Istvan es Szent Laszlo Korhaz-Rendelointeszet, Budapest
  - Bajcsy-Zsilinsky Korhaz, Budapest
  - Jasz-Nagykun-Szolnok Megyei, Szolnok
- Italy (7):
  - CRO Aviano, Aviano
  - A.O.U. Policlinico Vittorio Emanuele, Catania
  - A.O. Istituti Ospitalieri di Cremona, Cremona
  - A.O. Santa Croce e Carle Oespedale, Cuneo
  - Universita di Roma Sapienza, Rome
  - Azienda Ospedialiera Universitaria Senese, Siena
  - Oncologia medica Ospedale S. Vincenzo, Taormina
- Paula Stradina Kliniska Universitates slimnica, Riga, Latvia
- Lithuania (4):
  - Lithuanian University of Health Science Oncology Institute, Kaunas
  - Klaipeda University Hospital, Klaipėda
  - Vilnius University Hospital, Vilnius
  - National Cancer Institute, Vilnius
- Netherlands (7):
  - VU medical Center, Amsterdam
  - Wilhemina Ziekenhuis, Assen
  - Tergooi Ziekenhuizen, Hilversum
  - Spaarne Gasthuis, Hoofddorp
  - Oncology Medisch Centrum, Leeuwarden
  - UMC St.Radboud, Nijmegen
  - Oncology Maasstad Ziekenhuis, Rotterdam
- Poland (5):
  - Przychodnia Lekarska (KOMED), Konin
  - Szpital im M.Kopernika, Lodz
  - INSTYTUT im. Marii Sklodowskiej-Curie, Warsaw
  - Centrum Medyczne Ostrobramska, Warsaw
  - Akademicki Szpital Kliniczny im. Jana Mikulicza-Radeckiego, Wroclaw
- Portugal (3):
  - Hospital da Luz, Lisbon
  - Centro Hospitalar de Lisboa Norte, E.P.E - Hospital de Santa Maria, Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, E.P.E, Porto
- Serbia (4):
  - CHC Zemun, Belgrade
  - Clinical Center of Serbia, Belgrade
  - Institute of Oncology and Radiology of Serbia, Belgrade
  - KBC Bezanijska Kosa, Belgrade
- Slovakia (8):
  - J.Breza MEDICAL s.r.o., Bratislava
  - Urologicka ambulancia CUIMED s.r.o., Bratislava
  - Univerzitna nemocnica Martin, Martin
  - Urologicka ambulancia Uroexam, spol. s r.o., Nitra
  - UROX s.r.o., Piešťany
  - Urocentrum MILAB s.r.o., Prešov
  - Privatna urologicka ambulancia, Trenčín
  - Fakultna nemocnica s poliklinikou Zilina, Žilina
- Spain (10):
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranón, Madrid
  - Hosp. Clinico Univ. San Carlos, Madrid
  - Instituto de Investigaciones Sanitarias (IIS), Fundacíon Jimenez Díaz (FJD), Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncológico Clara Campal (CIOCC), Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Universitario Quiron Madrid, Pozuelo de Alarcón
- Sweden (2):
  - Örebro University Hospital, Örebrö
  - University Hospital Umeå, Dept Oncology, Umeå
- United Kingdom (9):
  - The Clatterbridge Cancer Centre, Bebington
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - St. Luke's Cancer Centre Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - Royal Free Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Northern Centre for Cancer Care, Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hensler M, Rakova J, Kasikova L, Lanickova T, Pasulka J, Holicek P, Hraska M, Hrnciarova T, Kadlecova P, Schoenenberger A, Sochorova K, Rozkova D, Sojka L, Drozenova J, Laco J, Horvath R, Podrazil M, Hongyan G, Brtnicky T, Halaska MJ, Rob L, Ryska A, Coosemans A, Vergote I, Garg AD, Cibula D, Bartunkova J, Spisek R, Fucikova J. Peripheral gene signatures reveal distinct cancer patient immunotypes with therapeutic implications for autologous DC-based vaccines. Oncoimmunology. 2022 Jul 22;11(1):2101596. doi: 10.1080/2162402X.2022.2101596. eCollection 2022. PMID 35898703
- [Derived] Vogelzang NJ, Beer TM, Gerritsen W, Oudard S, Wiechno P, Kukielka-Budny B, Samal V, Hajek J, Feyerabend S, Khoo V, Stenzl A, Csoszi T, Filipovic Z, Goncalves F, Prokhorov A, Cheung E, Hussain A, Sousa N, Bahl A, Hussain S, Fricke H, Kadlecova P, Scheiner T, Korolkiewicz RP, Bartunkova J, Spisek R; VIABLE Investigators. Efficacy and Safety of Autologous Dendritic Cell-Based Immunotherapy, Docetaxel, and Prednisone vs Placebo in Patients With Metastatic Castration-Resistant Prostate Cancer: The VIABLE Phase 3 Randomized Clinical Trial. JAMA Oncol. 2022 Apr 1;8(4):546-552. doi: 10.1001/jamaoncol.2021.7298. PMID 35142815

RESULTS

PARTICIPANT FLOW:
Groups:
- DCVAC/PCa With Standard of Care Chemotherapy: Combination therapy with dendritic cell vaccine for prostate cancer (DCVAC/PCa) and standard of care chemotherapy (docetaxel and prednisone)
Period: Overall Study
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Started | 787 | 395
Completed | 188 | 106
Not Completed | 599 | 289
Not completed — Protocol Violation | 2 | 0
Not completed — Unable to tolerate leukapheresis | 1 | 0
Not completed — Failure to produce study treatment | 6 | 0
Not completed — Death | 518 | 254
Not completed — Medical monitor's decision (active hepatitis B) | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 51 | 23
Not completed — Disease progression | 0 | 1
Not completed — Lost to Follow-up | 19 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy | Total
Number analyzed (Participants) | 787 | 395 | 1182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 272 | 107 | 379
  >=65 years | 515 | 288 | 803
Age, Continuous [Median (Full Range); unit: years] | 68.0 [46 to 89] | 69.0 [46 to 89] | 68.0 [46 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 787 | 395 | 1182
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 26 | 19 | 45
  White | 733 | 358 | 1091
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 18 | 11 | 29
Region of Enrollment [Number; unit: participants]
  Hungary | 28 | 14 | 42
  United States | 144 | 73 | 217
  Czechia | 102 | 40 | 142
  United Kingdom | 60 | 36 | 96
  Belarus | 13 | 18 | 31
  Portugal | 20 | 10 | 30
  Spain | 18 | 14 | 32
  Austria | 14 | 5 | 19
  Latvia | 0 | 2 | 2
  Netherlands | 29 | 19 | 48
  Sweden | 4 | 1 | 5
  Belgium | 20 | 11 | 31
  Denmark | 2 | 0 | 2
  Poland | 94 | 36 | 130
  Italy | 19 | 3 | 22
  Slovakia | 49 | 15 | 64
  Bulgaria | 15 | 10 | 25
  France | 18 | 12 | 30
  Lithuania | 6 | 5 | 11
  Serbia | 22 | 14 | 36
  Germany | 92 | 51 | 143
  Croatia | 18 | 6 | 24
Prostate-specific antigen [Median (Full Range); unit: ng/L] — Population: PSA available for 786 patients in the experimental arm (DCVAC/PCa) and 394 patients in the control arm (placebo)
  ng/L
    number analyzed (Participants) | 786 | 394 | 1180
    (all) | 46.35 [0.0 to 7500.0] | 54.02 [0.1 to 5000.0] | 47.87 [0.0 to 7500.0]

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival, Intention-to-treat Population
Description: Overall survival is defined as the time from randomization until death due to any cause.
Time Frame: From randomization to death due to any cause, up to 58 months
Population: Intention-to-treat population definition: All randomized patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 787 | 395
Months | 23.9 [21.6 to 25.3] | 24.3 [22.6 to 26.0]
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — Stratified by region (US vs other), prior abiraterone (Yes vs No), prior enzalutamide (Yes vs No) and Eastern Cooperative Oncology Group (ECOG) score (0, 1 vs 2); p = 0.596, Log Rank; Hazard Ratio (HR) = 1.042, 95% CI 2-sided [0.895 to 1.213]
Statistical Analysis 2: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Unstratified; Test type: Superiority; p = 0.648, Log Rank; Hazard Ratio (HR) = 1.036, 95% CI 2-sided [0.891 to 1.204]

2. Secondary Outcome: Overall Survival, Per Protocol Population
Description: Overall survival is defined as the time from randomization until death due to any cause.
Time Frame: From randomization to death due to any cause, up to 58 months
Population: Per protocol population definition:
  A subset of all randomized patients characterized by the following criteria:
  * had at least 1 post-baseline efficacy assessment
  * did not have any major protocol violation that would affect the endpoints being assessed
  * received at least 8 doses of DCVAC/PCa or placebo
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 438 | 284
Months | 29.7 [26.9 to 32.3] | 26.7 [24.7 to 28.8]
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — Stratified by region (US vs other), prior abiraterone (Yes vs No), prior enzalutamide (Yes vs No) and ECOG score (0, 1 vs 2); p = 0.335, Log Rank; Hazard Ratio (HR) = 0.908, 95% CI 2-sided [0.746 to 1.105]
Statistical Analysis 2: Comparison: DCVAC/PCa With Standard of Care Chemotherapy; Unstratified; Test type: Superiority; p = 0.192, Log Rank; Hazard Ratio (HR) = 0.879, 95% CI 2-sided [0.725 to 1.067]

3. Secondary Outcome: Overall Survival, Intention-to-treat Population, Abiraterone as Prior Therapy
Description: Overall survival is defined as the time from randomization until death due to any cause.
Time Frame: From randomization to death due to any cause, up to 58 months
Population: Intention-to-treat population definition: All randomized patients with abiraterone as prior therapy
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 187 | 103
Months | 16.6 [14.9 to 19.7] | 21.0 [16.6 to 24.1]
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — Stratified by region (US vs other), prior enzalutamide (Yes vs No) and ECOG score (0, 1 vs 2); p = 0.071, Log Rank; Hazard Ratio (HR) = 1.312, 95% CI 2-sided [0.976 to 1.762]
Statistical Analysis 2: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Unstratified; Test type: Superiority; p = 0.09, Log Rank; Hazard Ratio (HR) = 1.283, 95% CI 2-sided [0.961 to 1.712]

4. Secondary Outcome: Overall Survival, Intention-to-treat Population, Enzalutamide as Prior Therapy
Description: Overall survival is defined as the time from randomization until death due to any cause.
Time Frame: From randomization to death due to any cause, up to 58 months
Population: Intention-to-treat population definition: All randomized patients with enzalutamide as prior therapy
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 137 | 60
Months | 15.2 [13.3 to 18.3] | 21.4 [15.1 to 26.5]
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — Stratified by region (US vs other), prior abiraterone (Yes vs No) and ECOG score (0, 1 vs 2); p = 0.049, Log Rank; Hazard Ratio (HR) = 1.461, 95% CI 2-sided [1 to 2.134]
Statistical Analysis 2: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Unstratified; Test type: Superiority; p = 0.053, Log Rank; Hazard Ratio (HR) = 1.436, 95% CI 2-sided [0.993 to 2.077]

5. Secondary Outcome: Overall Survival, Intention-to-treat Population, no Prior Abiraterone or Enzalutamide
Description: Overall survival is defined as the time from randomization until death due to any cause.
Time Frame: From randomization to death due to any cause, up to 58 months
Population: Intention-to-treat population definition: All randomized patients with neither abiraterone nor enzalutamide as prior therapy
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 546 | 271
Months | 26.7 [25.2 to 28.8] | 25.7 [23.8 to 28.3]
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — Stratified by region (US vs other) and ECOG score (0, 1 vs 2); p = 0.501, Log Rank; Hazard Ratio (HR) = 0.938, 95% CI 2-sided [0.779 to 1.13]
Statistical Analysis 2: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Unstratified; Test type: Superiority; p = 0.512, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.781 to 1.131]

6. Secondary Outcome: Radiological Progression-free Survival, Intention-to-treat Population
Description: Progressive disease on bone scans was defined as a minimum of two new lesions. Visceral and nodal disease was evaluated according to RECIST 1.1 with modifications as described in the Statistical Analysis Plan.
Time Frame: Time from randomization to the date of the earliest objective evidence of either radiographic progression of bone lesions, radiographic progression of soft tissue lesions, or death due to any cause, up to 58 months
Population: Intention-to-treat population definition: All randomized patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 787 | 395
Months | 11.1 [11.0 to 11.4] | 11.1 [10.8 to 11.4]
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.886, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.863 to 1.136]
Statistical Analysis 2: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Unstratified; Test type: Superiority; p = 0.992, Log Rank; Hazard Ratio (HR) = 1.001, 95% CI 2-sided [0.875 to 1.145]

7. Secondary Outcome: Radiological Progression-free Survival, Per Protocol Population
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 438 | 284
Months | 11.2 [11.1 to 11.7] | 11.2 [11.0 to 11.8]
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.994, Log Rank; Hazard Ratio (HR) = 1.001, 95% CI 2-sided [0.847 to 1.184]
Statistical Analysis 2: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Unstratified; Test type: Superiority; p = 0.982, Log Rank; Hazard Ratio (HR) = 1.002, 95% CI 2-sided [0.851 to 1.18]

8. Secondary Outcome: Time to PSA Progression, Intention-to-treat Population
Description: The evidence of PSA progression is defined as: time from randomization to the date of PSA absolute increase ≥ 2 ng/mL and ≥ 25% above nadir or baseline values confirmed by a second consecutive value obtained at least 3 weeks later.
Time Frame: Time from randomization to the date of objective evidence of PSA progression (PSA absolute increase ≥ 2 ng/mL and ≥ 25% above nadir or baseline values providing confirmation by a second consecutive value obtained at least 3 weeks later), up to 39 months
Population: Intention-to-treat population definition: All randomized patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 787 | 395
Months | 10.5 [9.7 to 10.6] | 10.6 [10.4 to 10.7]
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.392, Log Rank; Hazard Ratio (HR) = 1.077, 95% CI 2-sided [0.909 to 1.277]
Statistical Analysis 2: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Unstratified; Test type: Superiority; p = 0.439, Log Rank; Hazard Ratio (HR) = 1.068, 95% CI 2-sided [0.905 to 1.262]

9. Secondary Outcome: Time to PSA Progression, Per Protocol Population
Description: as for outcome 8
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 438 | 284
Months | 10.5 [10.4 to 10.7] | 10.6 [10.4 to 10.7]
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.754, Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.857 to 1.238]
Statistical Analysis 2: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Unstratified; Test type: Superiority; p = 0.924, Log Rank; Hazard Ratio (HR) = 1.009, 95% CI 2-sided [0.844 to 1.207]

10. Secondary Outcome: Time to First Skeletal-related Event, Intention-to-treat Population
Description: Skeletal-related events included:
  * Radiation therapy to bone
  * Pathologic bone fracture
  * Spinal cord compression
  * Surgery to bone
  * Change in antineoplastic therapy to treat bone pain
Time Frame: Time from randomization to the date of the first skeletal-related event, up to 58 months
Population: Intention-to-treat population definition: All randomized patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 787 | 395
Months | NA [NA to NA] — Not reached; insufficient number of participants with events | NA [NA to NA] — Not reached; insufficient number of participants with events
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.732, Log Rank; Hazard Ratio (HR) = 0.918, 95% CI 2-sided [0.563 to 1.497]
Statistical Analysis 2: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Unstratified; Test type: Superiority; p = 0.713, Log Rank; Hazard Ratio (HR) = 0.913, 95% CI 2-sided [0.561 to 1.485]

11. Secondary Outcome: Time to First Skeletal-related Event, Per Protocol Population
Description: as for outcome 10
Time Frame: Time from randomization to the date of the first skeletal-related event, up to 58 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 438 | 284
Months | NA [NA to NA] — Not reached; insufficient number of participants with events | NA [NA to NA] — Not reached; insufficient number of participants with events
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.694, Log Rank; Hazard Ratio (HR) = 0.891, 95% CI 2-sided [0.5 to 1.587]
Statistical Analysis 2: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Unstratified; Test type: Superiority; p = 0.661, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.496 to 1.562]

12. Secondary Outcome: Time to Radiological Progression or Skeletal-related Event, Intention-to-treat Population
Description: Progressive disease on bone scans defined as a minimum of two new lesions. Visceral and nodal disease was evaluated according to RECIST 1.1 with modifications as described in the Statistical Analysis Plan.
  Skeletal-related events included:
  * Radiation therapy to bone
  * Pathologic bone fracture
  * Spinal cord compression
  * Surgery to bone
  * Change in antineoplastic therapy to treat bone pain
Time Frame: Time from randomization to the date of the first radiological progression or skeletal-related event, up to 58 months
Population: Intention-to-treat population definition: All randomized patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 787 | 395
Months | 11.1 [10.9 to 11.3] | 10.9 [10.5 to 11.2]
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.111, Log Rank; Hazard Ratio (HR) = 0.895, 95% CI 2-sided [0.781 to 1.027]
Statistical Analysis 2: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Unstratified; Test type: Superiority; p = 0.184, Log Rank; Hazard Ratio (HR) = 0.913, 95% CI 2-sided [0.798 to 1.044]

13. Secondary Outcome: Time to Radiological Progression or Skeletal-related Event, Per Protocol Population
Description: as for outcome 12
Time Frame: Time from randomization to the date of the first radiological progression or skeletal-related event, up to 58 months
Population: A subset of all randomized patients characterized by the following criteria:
  * had at least 1 post-baseline efficacy assessment
  * did not have any major protocol violation that would affect the endpoints being assessed
  * received at least 8 doses of DCVAC/PCa or placebo
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 438 | 284
Months | 11.1 [11.0 to 11.5] | 11.1 [10.8 to 11.3]
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.46, Log Rank; Hazard Ratio (HR) = 0.939, 95% CI 2-sided [0.795 to 1.11]
Statistical Analysis 2: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Unstratified; Test type: Superiority; p = 0.534, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.807 to 1.118]

14. Secondary Outcome: Proportion of Patients With Skeletal-related Events, Intention-to-treat Population
Description: as for outcome 12
Time Frame: From randomization to the end of the study, up to 57 months
Population: Intention-to-treat population definition: All randomized patients
Measure: Number; unit: Patients
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 787 | 395
Patients | 43 | 26
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — Adjusted by region (US vs other), prior abiraterone (Yes vs No), prior enzalutamide (Yes vs No) and ECOG score (0, 1 vs 2); p = 0.485, Log binomial model; Risk Ratio (RR) = 0.845, 95% CI 2-sided [0.528 to 1.355]

15. Secondary Outcome: Proportion of Patients With Skeletal-related Events, Per Protocol Population
Description: as for outcome 12
Time Frame: From randomization to the end of the study, up to 57 months
Population: as for outcome 13
Measure: Number; unit: Patients
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
Number analyzed (Participants) | 438 | 284
Patients | 28 | 20
Statistical Analysis 1: Comparison: DCVAC/PCa With Standard of Care Chemotherapy vs Placebo With Standard of Care Chemotherapy; Stratified; Test type: Superiority — [test comment as in outcome 14, analysis 1]; p = 0.768, Log binomial model; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.529 to 1.601]

ADVERSE EVENTS:
Time Frame: Up to 68 months. Adverse events (AEs) occurring after signing the informed consent until 30 days after the last dose of DCVAC/PCa or placebo were collected. Treatment-emergent AEs: Start date on or after the earliest start of chemotherapy or study treatment or adverse event worsened (increased in severity) on or after the earliest start of chemotherapy or study treatment. Deaths: From consent signature to study end.
Description: Mortality: in all randomized patients. AEs: in the safety population (received chemotherapy and/or at least 1 dose of DCVAC/PCa or placebo). At each contact, open-ended and non-leading verbal questioning of the patient by the investigator was used to inquire about AEs. Causal relationship of the AE to DCVAC/PCa or placebo was assessed by investigators. Disease progression-related events (as evaluated by investigators) were excluded from serious AE reporting but were captured as non-serious AEs.
Arm/Group | DCVAC/PCa With Standard of Care Chemotherapy | Placebo With Standard of Care Chemotherapy
All-Cause Mortality (participants affected / at risk) | 518/787 | 254/395
Serious Adverse Events (participants affected / at risk) | 237/749 | 150/379
Other Adverse Events (participants affected / at risk) | 670/749 | 365/379
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCVAC/PCa With Standard of Care Chemotherapy (N=749) | Placebo With Standard of Care Chemotherapy (N=379)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (5) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 2 (2) | 0 (0)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 3 (3) | 1 (1)
Catheter site inflammation (General disorders) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 5 (5) | 5 (5)
Fatigue (General disorders) | 5 (5) | 1 (1)
General physical health deterioration (General disorders) | 6 (6) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 9 (13) | 6 (9)
Sudden death (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 3 (4)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Computerised tomogram abnormal (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 7 (8) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 15 (15)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 9 (14) | 3 (3)
Bicytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 25 (27) | 29 (34)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 12 (12) | 5 (7)
Pancytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral venous thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Diabetic coma (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 2 (3)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 2 (2)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 2 (2) | 1 (1)
Superior sagittal sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 7 (8) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Vertigo CNS origin (Nervous system disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (6)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 4 (4)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 6 (8) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 6 (6) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal atrophy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 7 (8) | 4 (5)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0)
Abscess soft tissue (Infections and infestations) | 1 (2) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Catheter site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus oesophagitis (Infections and infestations) | 0 (0) | 1 (1)
Dermo-hypodermitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
Cholangitis infective (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Neutropenic sepsis (Infections and infestations) | 7 (7) | 5 (7)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0)
Paraspinal abscess (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 18 (18) | 11 (13)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 8 (8) | 5 (5)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 10 (13) | 8 (9)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 3 (3) | 0 (0)
Viral sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCVAC/PCa With Standard of Care Chemotherapy (N=749) | Placebo With Standard of Care Chemotherapy (N=379)
Hypertension (Vascular disorders) | 43 (56) | 34 (44)
Hypotension (Vascular disorders) | 40 (48) | 28 (39)
Asthenia (General disorders) | 106 (156) | 69 (107)
Fatigue (General disorders) | 268 (374) | 152 (219)
Mucosal inflammation (General disorders) | 28 (33) | 22 (37)
Oedema peripheral (General disorders) | 121 (146) | 87 (107)
Pyrexia (General disorders) | 76 (104) | 42 (64)
Insomnia (Psychiatric disorders) | 32 (33) | 24 (25)
Weight decreased (Investigations) | 46 (48) | 24 (25)
Anaemia (Blood and lymphatic system disorders) | 123 (159) | 76 (96)
Leukopenia (Blood and lymphatic system disorders) | 63 (103) | 33 (74)
Neutropenia (Blood and lymphatic system disorders) | 103 (177) | 54 (92)
Cough (Respiratory, thoracic and mediastinal disorders) | 82 (95) | 47 (54)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 82 (103) | 55 (65)
Dizziness (Nervous system disorders) | 41 (47) | 33 (40)
Dysgeusia (Nervous system disorders) | 80 (105) | 59 (91)
Headache (Nervous system disorders) | 35 (38) | 27 (33)
Hypoaesthesia (Nervous system disorders) | 32 (41) | 20 (25)
Neuropathy peripheral (Nervous system disorders) | 83 (110) | 54 (59)
Paraesthesia (Nervous system disorders) | 76 (95) | 33 (42)
Peripheral sensory neuropathy (Nervous system disorders) | 36 (39) | 28 (31)
Polyneuropathy (Nervous system disorders) | 44 (47) | 24 (28)
Taste disorder (Nervous system disorders) | 37 (39) | 21 (23)
Lacrimation increased (Eye disorders) | 29 (29) | 30 (32)
Abdominal pain (Gastrointestinal disorders) | 28 (31) | 23 (26)
Constipation (Gastrointestinal disorders) | 111 (133) | 71 (94)
Diarrhoea (Gastrointestinal disorders) | 204 (338) | 115 (183)
Dyspepsia (Gastrointestinal disorders) | 44 (47) | 22 (26)
Nausea (Gastrointestinal disorders) | 150 (196) | 96 (142)
Stomatitis (Gastrointestinal disorders) | 39 (54) | 24 (35)
Vomiting (Gastrointestinal disorders) | 78 (97) | 43 (53)
Alopecia (Skin and subcutaneous tissue disorders) | 222 (224) | 130 (131)
Nail disorder (Skin and subcutaneous tissue disorders) | 38 (41) | 28 (28)
Rash (Skin and subcutaneous tissue disorders) | 36 (40) | 22 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 114 (153) | 74 (110)
Back pain (Musculoskeletal and connective tissue disorders) | 113 (135) | 67 (79)
Bone pain (Musculoskeletal and connective tissue disorders) | 78 (91) | 26 (29)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 32 (36) | 23 (26)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 46 (51) | 24 (28)
Myalgia (Musculoskeletal and connective tissue disorders) | 53 (74) | 32 (47)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 87 (104) | 55 (74)
Decreased appetite (Metabolism and nutrition disorders) | 110 (137) | 79 (102)
Hyperglycaemia (Metabolism and nutrition disorders) | 56 (81) | 27 (41)
Nasopharyngitis (Infections and infestations) | 33 (39) | 22 (26)
Upper respiratory tract infection (Infections and infestations) | 34 (41) | 20 (23)
Urinary tract infection (Infections and infestations) | 53 (76) | 39 (66)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any formal publication of clinical trial results will be a collaborative effort between the sponsor and the investigator(s). All manuscripts or abstracts will be reviewed and approved in written by the sponsor before submission. The sponsor may request a delay in publication if there are important intellectual property concerns but does not have the right to suppress the publication of the clinical trial results indefinitely.

DOCUMENTS (2):
  • Study Protocol (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT02111577/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT02111577/SAP_001.pdf